CLINICAL TRIAL: NCT01034046
Title: Weight Loss and Visceral Fat Responses to Different Diet Compositions
Brief Title: Weight Loss and Abdominal Fat Responses to Different Diet Compositions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Jenny Craig, Inc. (Industry)
Responsible Party: Raymond Plodkowski, MD, University of Nevada School of Medicine, Reno
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B08/09-031
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2009-12

CONDITIONS: Obesity; Insulin Resistance; Metabolic Syndrome
Keywords: Obesity
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Sensitive Study Participants (Active Comparator): Insulin sensitive subjects stratified using fasting insulin levels.
  Interventions: Other: Low Carbohydrate Diet; Other: Low Fat Diet
- Insulin Resistant Study Subjects (Active Comparator): Insulin resistant subjects stratified using fasting insulin levels.
  Interventions: Other: Low Carbohydrate Diet; Other: Low Fat Diet

INTERVENTIONS:
Other: Low Carbohydrate Diet — Low carbohydrate diet (45% carbohydrate, 35% fat and 20% protein diet) administered utilizing meal replacements.
Other: Low Fat Diet — Low fat diet (60% carbohydrate, 20% fat and 20% protein diet) administered utilizing meal replacements.

SUMMARY:
The purpose of this study is to assess the effectiveness of two different reduced calorie diets that have different combinations of carbohydrate, fat, and protein content in 2 groups of study participants: insulin sensitive participants and insulin resistant participants. The hypothesis of the study is that people with high and low levels of insulin resistance may respond differently to different diet compositions in a real-world environment using meals that are commonly available.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 65 years of age.
* BMI 30-40 kg/m2
* Stable weight within 10 lb (+/-) for last 2 months

Exclusion Criteria:

* Pregnant or lactating.
* Must not currently be part of a structured weight loss program
* Taking a medication for diabetes (such as insulin, metformin, glyburide, glipizide, Byetta, pioglitazone, or rosiglitazone) or a medication such as systemic glucocorticoids that are known to affect blood sugar or blood insulin.
* Beck Depression Inventory (BDI Score >19 and/or positively endorses the suicide question on the BDI-II)
* Taking any chronic medication that has not had a stable dose for 1 month or longer.
* Diabetes mellitus defined as a fasting glucose ≥ 126 mg/dL on screening.
* Taking medications or dietary supplements that cause weight gain or weight loss (eg. antipsychotics (Seroquel, Zyprexa, and Risperdal) and/or anorectics).
* Clinically significant laboratory abnormalities at the opinion of the investigators.
* History of Bariatric Surgery
* A history of:

  * Type 2 diabetes, type 1 diabetes, or diabetes that is a result of pancreatic injury, or secondary forms of diabetes, e.g. Cushing's syndrome and acromegaly.
  * Liver disease, such as cirrhosis, or chronic active hepatitis B or C.
  * Use of investigational drugs within 30 days of visit 1
  * A pacemaker.
  * Hospitalization for depression in the past 6 months, history of moderate to severe major depression.
  * Any other condition that in the investigators' or sponsor's opinion could interfere with the results of the trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Change in weight in kg | 24 weeks

SECONDARY OUTCOMES:
Change in visceral fat via bioimpedance | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raymond A Plodkowski, MD, Principal Investigator — University of Nevada School of Medicine, Reno; Sachiko T St. Jeor, PhD, RD, Principal Investigator — University of Nevada School of Medicine, Reno
Locations (1):
- Center for Nutrition and Metabolism at the University of Nevada School of Medicine, Reno, Reno, Nevada, United States